CLINICAL TRIAL: NCT03985449
Title: Implementation of Uterine Fibroid Option Grid Patient Decision Aids Across Five Organizational Settings: a Randomized Stepped-wedge Study
Brief Title: Implementation of Uterine Fibroid Option Grid Patient Decision Aids Across Five Organizational Settings
Acronym: UPFRONT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other); Mayo Clinic (Other); Montefiore Medical Center (Other); Barnes-Jewish Hospital (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Glyn Jones-Elwyn, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: D19115
Record Dates: First submitted 2019-06-06; First posted 2019-06-13 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Uterine Fibroid
Keywords: Implementation; Shared decision making; Patient Decision Aids; Decision Support Intervention; Uterine Fibroids; Normalization Process Theory; Consolidated Framework for Implementation Research; Picture Superiority; Electronic Health Record; Coproduction
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Intervention Model Description: Stepped wedge trial with randomization at the clinic level. Patient enrollment will occur at five gynecology clinics in the United States. The uterine fibroid Option Grid patient decision aid intervention will be implemented in the 'active' implementation phase of the trial following a brief initiation session at each clinic to introduce clinicians to the intervention.
Masking Description: Data analysts will be blinded to the setting randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Implementation phase (Other): See the 'detailed description' section to read about the intervention(s) clinicians will use during the active implementation phase of the randomized stepped-wedge design.
  Interventions: Other: Uterine Fibroid Option Grid encounter patient decision aid (text only); Other: Uterine Fibroid Option Grid encounter patient decision aid (text + Pictures); Other: Uterine Fibroid Option Grid encounter patient decision aid (online)

INTERVENTIONS:
Other: Uterine Fibroid Option Grid encounter patient decision aid (text only) — The uterine fibroid Option Grid patient decision aid facilitates choice awareness and deliberation about treatment options when clinicians and patients discuss the management of uterine fibroids. The content is organized in a tabular format and is based on patients' frequently asked questions.
Other: Uterine Fibroid Option Grid encounter patient decision aid (text + Pictures) — The Picture Option Grid uses the same evidence as the text version while integrating images and simpler text, thus utilizing pictorial superiority to help patients better understand and remember information more easily compared to just using words.
Other: Uterine Fibroid Option Grid encounter patient decision aid (online) — Clinicians can click a link in the electronic health record that will lead them to the EBSCO Health website where they can click the treatment options relevant to the patient and generate a decision aid.

SUMMARY:
UPFRONT is a study that aims to use two implementation frameworks - the Consolidated Framework for Implementation Research and the Normalization Process Theory - to guide the implementation of a uterine fibroid patient decision aid, known as Option Grid, at five diverse gynecology settings across the United States. Option Grid provides evidence-based information on the various treatment options to help women across socioeconomic strata with symptomatic uterine fibroids make a preference-sensitive decision.

DETAILED DESCRIPTION:
Background & significance

Uterine fibroids are non-cancerous overgrowths of smooth muscle in the uterus. As they grow, a proportion of fibroids give rise to problems, such as heavy menstrual bleeding, pelvic pain, discomfort during sexual intercourse, and/or difficulty becoming pregnant. Some fibroids cause miscarriage, preterm birth, and increase the risk of cesarean birth. Multiple treatments are available: medication, removal of the inner layer of the uterus wall (endometrial ablation), removal of the uterus (hysterectomy) or part of the fibroid (myomectomy), or blocking some of the blood supply to the uterus (uterine artery embolization). Given the different consequences of treatment options, such as time away from work and impact on fertility, choosing the best option is sensitive to individual preferences. This study seeks to improve healthcare delivery and treatment choices for women of different socioeconomic status (SES) and health literacy levels experiencing symptoms from uterine fibroids.

Approximately 50% of women of reproductive age have fibroids, and at least 50% of these women have significant symptoms. These women report substantial impairment in quality of life and increased costs associated with the impact on daily living. While existing evidence is inconclusive about disparities in treatment choice, the associated socioeconomic burden is even greater in African-American women and those of lower SES. Despite a greater incidence and severity of symptomatic fibroids among African-American women, Hispanic women, and women of lower SES, one study shows that these women are less likely to undergo laparoscopic intervention, while another study found no significant differences between procedure rates between African-American and white women. Nevertheless, African-American women are more likely to experience poor treatment outcomes than white women.

A systematic review (2002) indicated that insufficient evidence exists about the comparative effectiveness of treatments for uterine fibroids. Viswanathan confirmed this view in 2007, saying that "the dearth of high-quality evidence is remarkable given how commonly this problem occurs." A report by Velentgas et al demonstrated similar outcomes between the uterine-sparing treatment options (endometrial ablation, uterine artery embolization, and myomectomy) on the onset of new or recurrent symptoms post-treatment. Myomectomy and uterine artery embolization led to a reduced risk of having a subsequent procedure compared to endometrial ablation. The lack of comparative evidence demonstrating superiority of any one treatment reinforces the role of shared decision making (SDM) in this context.

SDM is considered the pinnacle of patient-centered, ethical care and aims to promote two-way communication between clinicians and patients. Patient decision aids are interventions that provide evidence-based information to patients so they can make decisions that align with their preferences, thus facilitating the SDM process. For example, Option Grid encounter patient decision aids (ePDAs) are available in various formats (paper, picture, online interactive) and present information in a tabular format so patients can compare options. The use of Option Grids, and other similar ePDAs in other settings, also provide evidence that these tools are effective. A stepped-wedge study showed higher levels of SDM when Option Grid decision aids were used with patients who had knee osteoarthritis, as well as an increase in patient knowledge, without lengthening the encounter's duration. Similar results were found when Option Grid ePDAs were used by pediatricians with parents facing decisions about circumcision. In addition, five randomized trials using ePDAs at the Mayo Clinic, Rochester, Minnesota, have demonstrated their impact on SDM, whereas there is less evidence that PDAs used solely by patients before clinical encounters lead to observed changes in SDM.

The investigators have clear evidence from existing research and their own consultation with patient partners that women with fibroids wish to consider treatment trade-offs and engage in decision making processes. A trial of a pre-ePDA for women with uterine fibroids demonstrated impact on knowledge and satisfaction but no effect on concordance between preferences and decisions. A pre-post study by the current team has demonstrated that using the existing uterine fibroids Option Grid led to higher levels of SDM according to both observational and patient-reported measures. Despite interest among patients with uterine fibroids to participate in their healthcare decisions, and the positive impact of uterine fibroids ePDAs on SDM, implementation of SDM approaches in routine care remains challenging.

Implementation of SDM remains difficult across a range of healthcare settings, and success depends on more than simply distributing PDAs to patients. System and organizational barriers exist, related to incentives and established behavior patterns. There is evidence, however, that it is possible to implement SDM, particularly if it is supported by clinical champions, organizational strategies, and effective electronic medical record integration efforts, especially where tools fit well into workflows) and are useful with a diverse range of patients. The investigators searched for, but were unable to find, implementation studies of uterine fibroids ePDAs in clinical settings and conclude that a relevant gap exists.

To fill this gap, the investigators will use a multi-component SDM implementation strategy guided by the Consolidated Framework for Implementation Research and the Normalization Process Theory. The strategy includes: (1) assessment of organizational readiness for SDM using Measuring Organizational Readiness for patient Engagement (MORE) - a team-based survey to develop a tailored strategy at each site addressing potential organizational barriers to implementation; (2) online or in-person introduction to SDM and the Option Grid tools (this will include feedback and coaching); (3) clinician access to multiple formats of Option Grid ePDAs (text, picture, and online interactive version and printed Spanish versions), and; (4) the integration of a suggested SDM approach and new evidence (as appropriate) into existing clinical practice guidelines where feasible (e.g., the American College of Obstetricians and Gynecologists).

Study aims

The investigators propose to incorporate new comparative effectiveness evidence about uterine fibroid treatments into a multi-component SDM implementation strategy. The investigators will evaluate the impact of a multi-component SDM implementation strategy for the care of women who seek treatment for uterine fibroids at five diverse gynecology settings and across socioeconomic strata. The investigators will also examine the real-world clinical context from the five participating sites to determine the characteristics of a successfully (or not successfully) sustained a multi-component SDM strategy.

Study description

Procedure Prior to the pre-implementation phase, a minimum of 10 stakeholders from each site will complete the Measuring Organizational Readiness for patient Engagement (MORE) survey which is designed to measure a healthcare organization's willingness and ability to effectively implement patient engagement in healthcare. Participating clinicians will also complete the ADOPT survey to assess their attitudes toward patient decision aids at the start of the pre-implementation phase.

During the pre-implementation phase, eligible patients will be identified in advance by the project team at each project site through the sites' outpatient appointment systems. After their clinical encounter, clinic staff will provide eligible patients with a tablet computer to complete the consent form and fill out the survey. Patients will provide their email address in the survey so they can receive the follow-up survey three months post-encounter. To measure the extent to which clinicians involve patients in decision-making process, research assistants at each site will randomly audio-record five clinical encounters for each participating clinician.

The study interventions will be carefully described during a two-month initiation period for clinicians at participating sites, to occur between the pre- and active implementation periods.

Each site will decide which intervention (or a combination) they want to implement, as well as potentially suggest new ways of introducing the tool(s) to patients. This will be part of the implementation strategy and informed by the assessment of organizational readiness for patient engagement at each site completed during the pre-implementation phase. The study staff at each site will identify eligible patients ahead of their visits through their outpatient scheduling systems and will have the opportunity to mail or, where allowed by clinic policy, email the Option Grid before their appointment. Patients receiving the tools in advance would be instructed (with a cover letter) to use the tool to prepare for their encounter with their clinician. Patients will be encouraged to assess whether the frequently asked questions are issues that are also of concern to them, and to ask clinic staff to explain any parts which seem unclear to them.

The clinician will also have the option of presenting the Option Grid during the clinical encounter. To facilitate this process, the reception staff (or someone else in the clinic) could provide the tool to the patient before the visit just in case they did not bring their mailed copy. Or, the medical assistant can provide the tool to the patient upon rooming. The method of Option Grid presentation will be tailored to best fit the clinic flow at each site. Clinicians who have access to the online version of Option Grid will record use of the electronic tool into the patient's electronic medical record. Third, clinicians can give the Option Grid to the patient at the end of the encounter, so they can take it home and review its contents with others. This can be done by printing a paper copy, or if using the online version, by sending a URL link to the patient via email. Following the encounter, the patient will be provided with a tablet computer in order to provide consent and fill out the study surveys. Patients will be sent a follow-up link via email three months after the encounter to complete the follow-up survey. Like the pre-implementation phase, a research assistant at each site will audio-record five consecutive clinical encounters for each participating clinician to measure the extent to which clinicians involve patients in the decision-making process and complete the fidelity checklist.

To assess whether the intervention was sustainably implemented, the investigators will capture the perspective of professionals directly involved in the work of implementing complex interventions in healthcare using the NOMAD Normalization Process Theory instrument. The investigators will also assess clinician attitude using the ADOPT survey and conduct interviews with participating clinicians to determine the utility of the intervention, conduct a fidelity assessment, and calculate the percentage of eligible patients receiving the intervention. In addition, the investigators will have interview data which will help the investigators determine if systemic use is sustained.

ELIGIBILITY:
Inclusion Criteria:

* Patients showing new or recurrent symptoms of uterine fibroids (e.g. heavy menstrual bleeding, pelvic pressure or pain, etc.) who are seeking treatment.
* Assigned female sex at birth
* At least 18 years of age
* Speak English or Spanish
* Have the ability to complete short surveys online independently or assisted by a caregiver.

The investigators will also include health care professionals who will provide care to women with symptomatic uterine fibroids during the project duration at participating sites.

Exclusion Criteria:

* Patients who are under 18
* Patients not assigned female sex at birth
* Women who are postmenopausal because they will have different treatment options than the ones presented in this study's intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
The number of eligible patients that can be identified who receive the uterine fibroid Option Grid patient decision aid. | Month 1-14

SECONDARY OUTCOMES:
Measuring Organizational Readiness for patient Engagement (MORE) | Before week 1
  MORE is designed to measure a healthcare organization's willingness and ability to effectively implement patient engagement in healthcare. The measure contains 25 items each of which is scored on a four-point Likert-type scale (1=avoid/not important; 4=definitely involve/very important). Data from the measure will be analyzed to identify barriers and facilitators to implementation at each site.
Attitudes toward Decision Aids fOr PatienTs (ADOPT) | Month 1, Month 9, Month 22
  A measure of clinician attitudes to patient decision aids (PDA)s. Clinicians are asked to select one or more words that best describes their attitudes to the potential use of PDAs from a pool of ten words. It can be completed by clinicians who have, or have not, used PDAs.
Quality of shared decision making | Through Month 1-6, Month 8-14
  Observer OPTION-5 is a validated five-item scale, with each item rated from '0' to '4' where '0' represents absence of a shared decision making specific competency and '4' represents optimal performance.
Fidelity assessment | Through Month 10-14
  The fidelity assessment checklist enables the investigators to determine if an Option Grid was used, how and when it was delivered to the patient, whether or not the clinician made a treatment recommendation or elicited patient preference, and the identification of the final treatment decision. The checklist will help the investigators understand if the clinicians are using the tools as intended following initiation.
NoMAD Normalization Process Theory (NPT) survey | Month 6 and Month 22
  A 23-item instrument used for capturing the perspective of professionals who will be involved in implementing and using Option Grid in practice. The instrument contains four sections that ask questions on the various facets of implementing and using the intervention such as the effect that it has on workflow, the work and resources needed to drive implementation, and critical appraisal of the Option Grid, etc.
Utility of Option Grid patient decision aids and clinician approach to implementation | Month 14 and Month 22
  Semi-structured interviews, guided by the Normalization Process Theory, will be conducted with clinicians to assess the utility of the Option Grid tools and how they implemented the intervention in practice
Measuring shared decision making | Through Month 1-6, Month 8-14
  collaboRATE is a three-item, patient-reported experience measure of how patients perceive the effort that clinicians make to achieve three core aspects of shared decision making: informing patients, eliciting preferences, and integrating preferences into decisions made. Patients answer each question on a scale of 0 to 9. The measure is scored by using the percentage of patients who give the highest possible score of 9 for each item.
Uterine Fibroid Symptom and Health-Related Quality of Life Questionnaire (UFS-QOL) symptom severity subscale | Through Month 1-6, Month 8-14
  Patients will be asked to complete only the symptom severity subscale portion of the 37-item UFS-QOL questionnaire. The eight-item subscale asks patients how distressed their symptoms have made them feel over the past three months. Each item is scored on a Likert-type scale from '1' (None of the time) to '5' (All of the time).
The Comprehensive Score for financial Toxicity (COST) | Through Month 1-6, Month 8-14
  COST is a patient-reported outcome measure to assess financial toxicity in patients with cancer. The measure contains 11 items. Study stakeholders, including patient partners, felt that the majority of the items were not applicable for this study and wanted to minimize respondents' burden, so the investigators opted to only use 1 item. The questions reads: "I worry about the financial problems I will have in the future as a result of my illness or treatment", and the response scale is from '0' (not at all) to '4' (very much).
Chew Health Literacy Measure | Through Month 1-6, Month 8-14
  3-item validated measure of health literacy. The items are the following: How confident are you filling out medical forms by yourself? How often do you have someone (like a family member, friend, hospital/clinic worker, or caregiver) help you read hospital materials? How often do you have problems learning about your medical condition because of difficulty understanding written information? Patients who circle 'extremely' or 'quite a bit' on the Likert-type scale are considered to have high health literacy
Resource utilization (ambulatory and hospital) | Through Month 1-6, Month 8-14
  The follow-up survey will query eligible patients to self-report the number of outpatient (or visit to primary care clinician), inpatient, or emergency visits during the three-month follow-up period.
Treatment choice | Through Month 1-6, Month 8-14
  Patients will identify their intended treatment choice in the post-encounter survey. The investigators will also ask patients in the 3-month follow-up survey whether they have seen another clinician about another treatment, whether an Option Grid tool was used in that encounter, and to identify the final treatment option they selected.
Patient demographics | Through Month 1-6, Month 8-14
  The investigators will collect the patient's email address, health insurance status, age, race, gender, and spoken language via the survey they complete on the tablet computer post-encounter.

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Elwyn, MD, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
All patient survey data will be stored in a Qualtrics database, a HIPAA-compliant web-based data management system. The investigators will assign a unique study identification number to each member of the study team (including clinicians). All data including clinician demographic information (age, gender, and years of experience post-fellowship or year of residency) and the ADOPT, NoMAD and MORE survey responses will be stored in the Qualtrics database. All audio-recordings of clinical encounters and semi-structured interviews will be loaded by site-based project staff into Dartmouth's HIPAA-compliant SharePoint system that only the Dartmouth study team will be able to access. Each recording will be labeled with a unique identification number.

REFERENCES:
- [Background] Scalia P, Durand MA, Forcino RC, Schubbe D, Barr PJ, O'Brien N, O'Malley AJ, Foster T, Politi MC, Laughlin-Tommaso S, Banks E, Madden T, Anchan RM, Aarts JWM, Velentgas P, Balls-Berry J, Bacon C, Adams-Foster M, Mulligan CC, Venable S, Cochran NE, Elwyn G. Implementation of the uterine fibroids Option Grid patient decision aids across five organizational settings: a randomized stepped-wedge study protocol. Implement Sci. 2019 Sep 2;14(1):88. doi: 10.1186/s13012-019-0933-z. PMID 31477140
- [Derived] Forcino RC, Durand MA, Schubbe D, Engel J, Banks E, Laughlin-Tommaso SK, Foster T, Madden T, Anchan RM, Politi M, Lindholm A, Gargiulo RM, Seshan M, Tomaino M, Zhang J, Acquilano SC, Akinfe S, Sharma A, Aarts JWM, Elwyn G. The UPFRONT project: tailored implementation and evaluation of a patient decision aid to support shared decision-making about management of symptomatic uterine fibroids. Implement Sci. 2024 Nov 5;19(1):75. doi: 10.1186/s13012-024-01404-5. PMID 39501337
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31477140/